CLINICAL TRIAL: NCT00112619
Title: A Phase I Pharmacokinetic Optimal Dosing Study of Intraventricular Topotecan for Children With Neoplastic Meningitis
Brief Title: Topotecan in Treating Young Patients With Neoplastic Meningitis Due to Leukemia, Lymphoma, or Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual and company withdrawing support to supply the drug
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett, Executive Director Operations and Biostatistics Center, Pediatric Brain Tumor Consortium
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000430504; U01CA081457 (NIH); PBTC-019
Record Dates: First submitted 2005-06-02; First posted 2005-06-03 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Brain and Central Nervous System Tumors; Carcinoma of Unknown Primary; Leukemia; Lymphoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; unspecified childhood solid tumor, protocol specific; childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebral astrocytoma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; recurrent childhood ependymoma; recurrent childhood medulloblastoma; childhood oligodendroglioma; recurrent childhood supratentorial primitive neuroectodermal tumor; leptomeningeal metastases; recurrent carcinoma of unknown primary; childhood central nervous system germ cell tumor; childhood chronic myelogenous leukemia; juvenile myelomonocytic leukemia; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood visual pathway and hypothalamic glioma; childhood atypical teratoid/rhabdoid tumor; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; relapsing chronic myelogenous leukemia; recurrent childhood pineoblastoma; recurrent childhood subependymal giant cell astrocytoma; meningeal leukemia; secondary central nervous system Hodgkin lymphoma; secondary central nervous system non-Hodgkin lymphoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasms, Unknown Primary; Leukemia; Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Astrocytoma; Choroid Plexus Neoplasms; Familial ependymoma; Medulloblastoma; Oligodendroglioma; Meningeal Carcinomatosis; Leukemia, Myelomonocytic, Juvenile; Recurrence; Optic Nerve Glioma; Rhabdoid Tumor | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: topotecan hydrochloride — Participants receive intraventricular topotecan, .2 mg, administered via an indwelling ventricular reservoir daily for 5 consecutive days during weeks 1 and 3 of the first four weeks of therapy (induction), during weeks 5 and 8 of the next 6 weeks of therapy (consolidation), and during weeks 11, 15, 19, 23, 27, 31, 35, 39, 43, 47, and 51 (maintenance therapy).
  Other Names: Hycamptin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects, best way to give, and best dose of topotecan when given by intraventricular infusion in treating young patients with neoplastic meningitis due to leukemia, lymphoma, or solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose (MTD) of intraventricular topotecan in young patients with neoplastic meningitis secondary to leukemia, lymphoma, or solid tumors.
* Determine the toxic effects and dose-limiting toxicity of this drug in these patients.
* Determine whether the MTD of this drug is also the pharmacokinetic optimal dose, defined by the topotecan lactone concentration in the cerebral spinal fluid (CSF), in these patients.

Secondary

* Determine, preliminarily, the antitumor activity of this drug in these patients.
* Determine the pharmacokinetics of this drug in the CSF of these patients.
* Correlate observed effects of post-treatment central review imaging (if feasible) with response to this drug in these patients.

OUTLINE: This is a non-randomized, dose-escalation, multicenter study.

* Induction therapy (weeks 1-4): Patients receive topotecan intraventricularly* over 5 minutes on days 1-5 in weeks 1 and 3. Patients then proceed to consolidation therapy in week 5.

NOTE: *Patients who are willing, receive 1 intralumbar (instead of intraventricular) dose of topotecan on day 1 of week 3 only.

* Consolidation therapy (weeks 5-10): Patients receive topotecan intraventricularly on days 1-5 in weeks 5 and 8. Patients then proceed to maintenance therapy in week 11.
* Maintenance therapy (weeks 11-54): Patients receive topotecan intraventricularly on days 1-5 in weeks 11, 15, 19, 23, 27, 31, 35, 39, 43, 47, and 51.

Cohorts of 3-6 patients receive escalating doses of intraventricular topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Once the MTD is determined, the cohort is expanded to 25 patients and the MTD is declared the pharmacokinetic optimal dose provided 23 of 25 patients treated at the MTD achieve the target pharmacokinetic parameter.

PROJECTED ACCRUAL: A total of 28-49 patients will be accrued for this study within 9-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neoplastic meningitis secondary to leukemia, lymphoma (including AIDS-related lymphoma), or solid tumor (including primary CNS tumors or carcinomas of unknown primary site), defined by 1 of the following criteria:

  * Cerebral spinal fluid (CSF) cell count > 5/μL AND evidence of blast cells on cytospin or by cytology (for patients with leukemia or lymphoma)
  * Presence of tumor cells on cytospin or cytology OR unequivocal presence of meningeal disease by MRI (for patients with solid tumor)
* No conventional therapy for neoplastic meningitis exists

  * Patients with CNS leukemia or lymphoma must be refractory to conventional therapy, including radiotherapy (i.e., second or greater relapse)
* Patients with CNS leukemia or lymphoma must have had a negative bone marrow aspiration within the past 2 weeks
* No clinical evidence of obstructive hydrocephalus
* No compartmentalization of CSF flow by radioisotope indium In 111 or technetium Tc 99 DTPA flow study
* No ventriculoperitoneal or ventriculoatrial shunt unless patient is completely shunt-independent
* No impending spinal cord compression or other CNS involvement (e.g., acute visual loss secondary to optic nerve involvement) requiring emergent local radiotherapy

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Lansky 60-100% (≤ 16 years of age) OR
* Karnofsky 60-100% (> 16 years of age)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Calcium ≥ 7 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Sodium 125-150 mmol/L
* Magnesium ≥ 0.7 mmol/L
* Must have or be willing to have an intraventricular access device (i.e., Ommaya reservoir)
* No uncontrolled infection

  * HIV-positive patients with AIDS-related lymphomatous meningitis are eligible
* No other significant uncontrolled systemic medical illness that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior biologic therapy or immunotherapy

Chemotherapy

* Recovered from prior chemotherapy
* At least 1 week since prior intra-colony stimulating factory (CSF) chemotherapy (2 weeks for liposomal cytarabine)
* At least 3 weeks since prior systemic chemotherapy for leptomeningeal disease
* Concurrent systemic chemotherapy to control systemic disease or bulk CNS disease allowed provided the systemic chemotherapy is not an investigational agent OR any of the following:

  * High-dose (> 1 g/m^2) methotrexate
  * High-dose (> 1 g/m^2) cytarabine
  * Fluorouracil
  * Capecitabine
  * Thiotepa
  * Nitrosoureas
  * Topotecan

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* At least 8 weeks since prior craniospinal radiotherapy and recovered
* No concurrent CNS radiotherapy

  * Concurrent radiotherapy to extra-CNS sites (e.g., painful bone metastases not in the craniospinal axis) allowed

Surgery

* Not specified

Other

* More than 2 weeks since prior and no other concurrent investigational agents
* No other concurrent intra-CSF or systemic therapy for leptomeningeal disease

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Estimate the maximum tolerated dose of intraventricular topotecan on this schedule | First 14 days of therapy
Number of patients with dose-limiting toxicity | First 14 days of therapy
Estimate the dose of intraventricular topotecan that will result in cerebrospinal fluid lactone concentrations exceeding 1 ng/mL for at least 8 hours after an intrathecal injection | Day 1 of Week 1

SECONDARY OUTCOMES:
Number of patients with objective documentation of tumor response to intraventricular topotecan | Weeks 5, 11 and then every 12 weeks until off study
  MRI of the brain and spine is obtained pre-consolidation, pre-maintenance, and then every 12 weeks in maintenance.
Pharmacokinetics | Day 1 of Week 1
  The cerebrospinal fluid (CSF) concentration-time profile for topotecan after intrathecal CSF administration will be modeled from the CSF samples collected on day 1 of week 1. Individual pharmacokinetic parameters estimated will include volume of central compartment, elimination rate constant, half-life, and clearance.
Correlation of imaging parameters with tumor response | Pre-treatment, week 5, week 11, and then every 12 weeks until off study
  MRI scans of the brain and spine is obtained pre-treament, pre-consolidation, pre-maintenance, and then every 12 weeks on maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Susan M. Blaney, MD, Study Chair — Baylor College of Medicine
Locations (11):
- United States (11):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Dan L. Duncan Cancer Center at Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington